CLINICAL TRIAL: NCT01452594
Title: Analysis of Immune Reactions Occurring in Normal Volunteers Upon Administration of the Topical Immunomodulator Diphenylcyclopropenone
Brief Title: Analysis of Diphenylcyclopropenone (DPCP) in Normals
Status: Completed | Type: Observational
Sponsor: Rockefeller University (Other)
Responsible Party: Principal Investigator, Nicholas Gulati, Biomedical Fellow, Rockefeller University
Other Study IDs: JKR-0742
Record Dates: First submitted 2011-10-12; First posted 2011-10-17 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — diphenylcyclopropenone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin Biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diphenylcyclopropenone: topical gel administration to skin
  Interventions: Drug: Diphenylcyclopropenone; Drug: Placebo

INTERVENTIONS:
Drug: Diphenylcyclopropenone — Topical administration
Drug: Placebo — Placebo

SUMMARY:
The drug diphenylcyclopropenone, or DPCP, modifies the immune system and has been shown to be effective in treating certain kinds of cancer. This study hopes to improve our understanding of how this drug helps create an effective immune response.

DETAILED DESCRIPTION:
The immune system is the primary line of defense against infections and other things perceived as foreign to the body. Unfortunately, this immune system often fails to eliminate tumors or other cancerous growths. The drug diphenylcyclopropenone, or DPCP, modifies the immune system and has been shown to be effective in treating certain kinds of cancer. This study hopes to improve our understanding of how this drug helps create an effective immune response. In order to reach this goal, normal volunteers will be given the DPCP drug in the form of a gel or a placebo gel (gel without the active chemical) on a few small areas of skin. Then, biopsies will be taken of the skin at the sites where the active drug was placed. Also, small biopsies will be taken from opposite areas of skin which received placebo gel to serve as controls. The biopsied skin samples will then be studied by methods such as immunohistochemistry and microarray analysis which will help define the immune reaction caused by DPCP. The rationale for the study is to better understand how the immune system can be activated to produce cells that may fight infections or cancers.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female between 18 and 60 years of age
* Able to give verbal and written informed consent
* For women of childbearing potential (WOCBP) or in men whose partners may become pregnant, willingness to use an acceptable method of contraception to prevent pregnancy for the duration of the study (while receiving study medication and for one month following the last dose of study medication). Acceptable forms of contraception are listed in the protocol.
* Must have a negative urine pregnancy test (for WOCBP)

Exclusion Criteria:

* Subjects taking any of the following systemic or topical therapies within 4 weeks of enrollment: corticosteroids, immunosuppressants, and/or any other medications that may affect the outcome of the study
* Known sensitivity to bandage or adhesive tape.
* Subjects who have active localized or systemic medical conditions that, in the opinion of the investigator, would preclude or make unsafe their participation in the study
* Subjects with any underlying concomitant diagnosis that may influence immune reactions (e.g. eczema, psoriasis, lupus)
* Subjects who are nursing mothers, pregnant, or planning to become pregnant at anytime during the course of the study or within 30 days of study completion
* Subjects who are unable to comply with study procedures, communicate effectively, cooperate with the investigator, or are unable to understand the study
* Subjects who have been treated with another investigational device or drug within 30 days of enrollment
* HIV positive as determined by self-reported history and/or a HIV POCT at screening
* History, physical, social or lab findings suggestive of any medical or psychological condition that would, in the opinion of the PI, make the candidate ineligible for the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Volunteers
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Krueger, MD,PhD, Principal Investigator — Rockefeller University
Locations (1):
- The Rockefeller University, New York, New York, United States